CLINICAL TRIAL: NCT00079300
Title: Double-Blind, Vehicle-Controlled Study to Evaluate Apoptosis in Basal Cell Carcinoma Treated With Aldara™ (Imiquimod) Cream, 5% Applied Once or Twice a Day
Brief Title: Imiquimod Cream in Treating Patients With Basal Cell Skin Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Naval Medical Center (U.S. Federal Agency)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000355151; NCI-02-CC-0289; 3M-1454-IMIQ; NCT00045851 (obsolete NCT alias)
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Non-melanomatous Skin Cancer
Keywords: basal cell carcinoma of the skin
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Imiquimod

INTERVENTIONS:
Drug: imiquimod
Procedure: conventional surgery

SUMMARY:
RATIONALE: Biological therapies, such as imiquimod cream, work in different ways to stimulate the immune system and stop tumor cells from growing.

PURPOSE: This randomized phase I trial is studying how well imiquimod cream works in treating patients with basal cell skin cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare levels of apoptosis in patients with basal cell skin cancer treated with vs without imiquimod 5% cream.

Secondary

* Compare levels of apoptosis in patients treated with this drug on two different administration schedules.

OUTLINE: This is a randomized, double-blind, placebo-controlled, parallel-group study.

Patients undergo fine needle aspiration and punch biopsies of the target lesion. Patients are then randomized to 1 of 8 treatment arms and begin therapy within 30 days after biopsy.

* Arm I: Patients apply topical imiquimod to the target lesion once every 12 hours on days 1 and 2 for a total of 4 doses.
* Arm II: Patients apply topical placebo to the target lesion once every 12 hours on days 1 and 2 for a total of 4 doses.
* Arm III: Patients apply topical imiquimod to the target lesion once every 24 hours on days 1-4 for a total of 4 doses.
* Arm IV: Patients apply topical placebo to the target lesion once every 24 hours on days 1-4 for a total of 4 doses.
* Arm V: Patients apply topical imiquimod to the target lesion once every 12 hours on days 1-4 for a total of 8 doses.
* Arm VI: Patients apply topical placebo to the target lesion once every 12 hours on days 1-4 for a total of 8 doses.
* Arm VII: Patients apply topical imiquimod to the target lesion once every 24 hours on days 1-8 for a total of 8 doses.
* Arm VIII: Patients apply topical placebo to the target lesion every 24 hours on days 1-8 for a total of 8 doses.

All patients undergo excision of the target tumor within 18-30 hours after the last topical treatment.

Patients are followed at 7-14 days.

PROJECTED ACCRUAL: A total of 48 patients (8 per treatment arm and 4 per placebo arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed basal cell skin cancer

  * Superficial or nodular disease
  * No aggressive disease
* At least 1 lesion at least 7 mm in diameter that meets the following criteria:

  * Primary tumor (no recurrent or previously treated disease)
  * Located on the scalp, face (including ears), trunk, or proximal extremities
  * Qualifies for surgical excision as primary therapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No evidence of a clinically significant or unstable medical condition that would adversely affect blood circulation

Other

* No dermatological disease (e.g., psoriasis or eczema) at the treatment site that may be exacerbated by treatment with imiquimod or interfere with examination
* No febrile viral infection within the past 4 weeks
* No evidence of a clinically significant or unstable medical condition that would adversely affect immune function

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior interferon, interferon inducers, or immunomodulators
* No concurrent interferon, interferon inducers, or immunomodulators

Chemotherapy

* More than 6 months since prior anticancer chemotherapy
* No concurrent anticancer chemotherapy

Endocrine therapy

* More than 4 weeks since prior oral or inhaled (more than 600 mcg/day for fluticasone or equivalent) corticosteroids
* More than 4 weeks since prior topical steroids to the target tumor
* Concurrent topical steroids in non-target areas are allowed provided amount used is ≤ 2 g of fluorinated steroids daily for > 1 week or 6 g of beclomethasone for > 1 week
* No concurrent oral or inhaled corticosteroids

Radiotherapy

* Not specified

Surgery

* More than 4 months since prior biopsy

Other

* More than 4 weeks since prior immunosuppressive therapies
* More than 4 weeks since prior cytotoxic or investigational drugs
* No concurrent immunosuppressive therapies
* No other concurrent cytotoxic or investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco M. Marincola, MD, Principal Investigator — NIH - Warren Grant Magnuson Clinical Center
Locations (1):
- NIH - Warren Grant Magnuson Clinical Center, Bethesda, Maryland, United States